CLINICAL TRIAL: NCT07164937
Title: Advanced Imaging and Multimodal Posture and Gait Analysis in Patients Affected by Facio-scapulo-humeral Dystrophy (FSHD): Development of an Innovative Model for Orthopedic Device Design
Brief Title: Imaging and Gait Analysis in FSHD Patients
Acronym: FSH-3DGait
Status: Enrolling by invitation | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6687
Record Dates: First submitted 2024-11-21; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-09

CONDITIONS: FSHD - Facioscapulohumeral Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Facioscapulohumeral muscular dystrophy (FSHD) is a common genetic muscle disorder characterized by progressive and often asymmetric muscle weakness, with high variability in clinical severity and disease progression. This study aims to integrate advanced imaging and motion analysis technologies to comprehensively evaluate the impact of FSHD on muscle degeneration and motor functionality.

The primary objective is to characterize the distribution and severity of muscle degeneration using magnetic resonance imaging (MRI) and correlate these findings with motor functionality profiles in a cohort of FSHD patients.

Secondary objectives include:

Describing gait and posture through the analysis of functional parameters using 3D-motion capture technologies.

Quantifying changes in gait and posture parameters before and after personalized orthopedic interventions, assessed with functional clinical scales and 3D-motion capture analysis.

This single-center, observational study will recruit 40 genetically confirmed FSHD patients from routine clinical follow-ups at the Policlinico Gemelli. Patients will undergo MRI to assess the degree of muscle fatty replacement (T1-score) and 3D Gait Analysis to capture biomechanical parameters such as kinematics, ground reaction forces, and muscle activation. Functional assessments will include tests like the Six-Minute Walk Test (6MWT) and Timed Up & Go Test (TUG), alongside standardized scales for balance, fatigue, pain, and quality of life.

The study seeks to identify novel clinical and biomechanical outcome measures that can stratify FSHD patients and evaluate therapeutic interventions. By correlating MRI patterns with motor deficits and analyzing the impact of orthopedic devices, the study aims to inform personalized rehabilitation strategies and support the design of clinical trials.

DETAILED DESCRIPTION:
Facioscapulohumeral muscular dystrophy (FSHD) is a common hereditary myopathy characterized by asymmetric involvement of facial, scapular, truncal, and lower limb muscles. Disease progression is highly variable, ranging from mild weakness to severe motor disability. Although muscle MRI has emerged as a sensitive tool to detect fatty replacement and disease activity, its integration with quantitative functional assessments is still limited.

This study is designed to explore the relationship between structural changes observed on MRI and functional motor performance in a cohort of adult FSHD patients. By combining whole-body MRI with standardized clinical evaluations and advanced 3D motion analysis, the project aims to provide a multidimensional characterization of motor impairment in FSHD.

The protocol foresees the acquisition of MRI scans and gait analysis data within a defined temporal window, ensuring comparability of structural and functional information. MRI data will be analyzed to derive a semiquantitative T1-score reflecting the burden of fatty infiltration, as well as STIR sequences for signs of muscle inflammation. These imaging findings will then be correlated with clinical outcome measures, including validated severity scales, timed functional tests, and motion capture-derived biomechanical parameters.

An additional exploratory component concerns the assessment of personalized orthopedic interventions, with pre- and post-application gait analysis sessions. This approach will allow the evaluation of the short-term functional impact of targeted assistive devices, generating insights for individualized rehabilitation strategies.

The expected contribution of this study is twofold: first, to validate MRI-based biomarkers and biomechanical metrics as reliable outcome measures for FSHD; and second, to establish an integrated framework for assessing motor impairment that may be applied in future interventional trials and in routine clinical management.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years. Genetically confirmed diagnosis of Facioscapulohumeral Muscular Dystrophy (FSHD).

Availability of:

Muscle MRI images. 3D Gait Analysis data (with or without personalized orthopedic aids). Both MRI and Gait Analysis performed within a maximum interval of 6 months from each other.

Regular neurological follow-ups as part of routine clinical care. Signed informed consent for participation in the study.

Exclusion Criteria:

* Age < 18 years.

Unavailability of:

Muscle MRI images. 3D Gait Analysis data performed within a maximum interval of 6 months from each other.

Refusal or inability to provide signed informed consent for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by FSHD
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Global T1-score and Regional T1-score Correlation: | At the enrollement
  Evaluation of the global T1-score and individual regional T1-scores (neck, shoulder girdle, trunk, pelvis, and lower limbs) derived from MRI ( minimun T1 score 0= normal; maximum T1 score 4= completely involved).
  Correlation of these scores with motor functionality parameters, including demographic data, clinical severity scales, functional clinical scales, and biomechanical parameters from 3D Gait Analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Enzo Ricci, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- UOC Neurologia, Rome, Italy